CLINICAL TRIAL: NCT00395668
Title: Assessment of Acute Changes in Cognitive Performance Arising From Exposure to TETRA Handset.
Brief Title: TETRA (Terrestrial Trunked Radio)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other); Aarhus University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2103-05-0005; Project nr. 0501- (Dept. ID)
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Cognitive Performance; Well-Being
Keywords: TETRA; EMF; Human exposure study; Symptoms; Well-being; Cognitive function

INTERVENTIONS:
Device: TETRA (at lowest carrier freq, std TDMA pulse at 17,6 Hz).

SUMMARY:
The purpose of this study is to investigate if electromagnetic radiation from TETRA handset can influence cognitive function and the well-being of healthy adults. Furthermore, the purpose is to provide any special information about the subjects which can cause the possible reactions.

DETAILED DESCRIPTION:
TETRA is the term used to describe the technology known as Terrestrial Trunked Radio. It is the European standard digital mobile radio communication system. TETRA has primarily been developed to enable the deployment of secure, digital PMR (Professional Mobile Radio) services required by the public safety and emergency services (police, fire and paramedics). The TETRA system is specified to work within the VHF and UHF bands (150 MHz to 900 MHz) [Chadwick, 2003], and operates most often at frequencies around 400 MHz. The lower frequency means that TETRA is less vulnerable to interference, which is a vital aspect of communications for the emergency services. The system makes it possible to offer complete coverage for the emergency services. One of the TETRA features is that the signal is transmitted in bursts that repeat. The result is a power modulation of some of the RF signal at a frequency of 17,6 Hz (times pr. second) [NRPB, 2001]. This pulsing has led to concerns about its effect on health. Since this pulsing only occurs for transmission from TETRA handset and not from the base stations, most concerns is related to the health effect on the users of TETRA handset.

The aim is to asses whether exposure to TETRA handset can affect cognitive functions and high level brain functions such as learning and problem solving the volunteers will be tested by comparing performance with and without exposure. Sham exposure (no radiation from the handset) vs. TETRA signal (at the lowest carrier frequency, standard TDMA pulsing at 17,6 Hz and a selection of lengths of exposures at the realistic SAR value).

56 healthy males aged 25-50 year working within public safety and emergency services (police, fire and paramedics), is planned to be used in this study. Subjects must be identified as potential users of the TETRA system.

A climatic chamber at the Department of Environmental and Occupational Medicine, Aarhus University, is modified with absorbing lining to dampen reflections from the walls. The climatic chamber is modified to make it a screened room to prevent external RF fields, and to some extent low frequency fields, to enter the chamber. Except for cables to the keyboard and screen there are no other electromagnetic radiators in the chamber. The study will be double blinded as any noise (acoustic and electric) related to exposure will be the same and the person responsible for exposure and exposure assessment will not be able to see each other. The only investigator knowledgeable about the exposure will have no contact with subjects and staff doing measurement. This double blinding will continue until the basic statistical analyses have been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age 25-50
* Males
* Right-handers

Exclusion Criteria:

* Subjects with current or previous cardiovascular disease
* Subjects with current or previous fractured scull
* Subjects with diseases, which could involve a risk for the subject or possible influence the outcome measurements

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2006-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary analysis is the comparison
of the placebo exposure (no radiation) and the TETRA signal
The primary outcome for this analysis is the Trail Making B (time in seconds).

SECONDARY OUTCOMES:
Reaction Time (RTI), complex reaction and movement time
Digit Span forward and backward
'Headache' and 'concentration difficulties' (VAS-scale)

CONTACTS AND LOCATIONS:
Overall Officials: Søren K. Kjærgaard, Ass.Prof.PhD, Principal Investigator — Institute of Public Health, University of Aarhus, Vennelyst Boulevard 6, Build. 1260
Locations (1):
- Dept. of Environmental and Occupational Medicine, Institute of Public Health, University of Aarhus, Vennelyst Boulevard 6, Build. 1260, Aarhus C, Denmark